CLINICAL TRIAL: NCT05434481
Title: MITAORTA - Role of Mitochondrial Dynamic in Aneurysm and Dissection of Ascending Thoracic Aorta
Acronym: MITAORTA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Collaborators: Fondation de l'Avenir (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2022-A00719-34
Record Dates: First submitted 2022-06-03; First posted 2022-06-28 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Aortic Aneurysm and Dissection
Keywords: extracellular matrix; cell survival; oxydative stress; mitochondrial fusion; metabolomic profiling of aortic aneurym; metabolomic profilng of aortic dissection
MeSH Terms: conditions — Aortic Dissection

STUDY DESIGN:
Intervention Model Description: Aneurysm and Dissection of Ascending Thoracic Aorta
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Aneurysm group (Active Comparator): Patients operated for aneurysm of the ascending aorta according the guidelines on the diagnosis and treatment of aortic diseases (European Society of Cardiology - 2014).
  Interventions: Other: Mitochondrial dynamic analysis in the aorta samples and metabolomic profiling in the aortic diseases
- Type A aortic dissection group (Active Comparator): Patients operated for type A aortic dissection according the guidelines on the diagnosis and treatment of aortic diseases (European Society of Cardiology - 2014).
  Interventions: Other: Mitochondrial dynamic analysis in the aorta samples and metabolomic profiling in the aortic diseases
- Control group (Sham Comparator): Patients without aortic aneurysm or aortic dissection operated for aortic valve replacement (AVR) and/or coronary artery bypass with a saphenous vein graft for proximal aortic anastomosis to collect the aortic sample. For patients operated for AVR, an aortic sample will be collected before closing the aorta.
  Interventions: Other: Mitochondrial dynamic analysis in the aorta samples and metabolomic profiling in the aortic diseases

INTERVENTIONS:
Other: Mitochondrial dynamic analysis in the aorta samples and metabolomic profiling in the aortic diseases — * For each patient: a segment of aorta will be sampled and cutted into 4 parts
    * 1 fragment placed in a Falcon tube containing DMEM (Dulbecco's Modified Eagle Medium, Thermo Fisher®), temporarily stored at + 4°C, for primary culture of smooth muscle cells will allow analysis of the mitochondrial network.
    * 1 fragment placed in a Falcon tube containing Allprotect Tissue Reagent (QIAGEN®), stored at -80°C for gene (RT-PCR) and protein (Western Blot) analysis.
    * 2 fragments each placed in dry cryotube stored at - 80°C will be used for metabolomic analysis.
  * For each patient, 2 arterial blood samples will be collected before general anaesthesia
    * One tube of whole blood stored at -80°C for metabolomic analysis.
    * One tube of blood stored at -80°C for plasma cytokines

SUMMARY:
The main objective is to compare the mitochondrial dynamic between patients operated for aneurysm of ascending aorta or type A aortic dissection (AAD) or control group

DETAILED DESCRIPTION:
In an aortic aneurysm process, the alteration of the extracellular matrix (ECM) as well as the apoptosis of the smooth muscle cells are due to inflammatory phenomena and oxydative stress, involving mitochondria which has a key place within cells.

Mitochondrial fusion and fission constitute mitochondrial dynamic and are involved in the mechanisms described above.

The alteration of mitochondrial dynamics has been demonstrated in many pathologies, in particular neurological, cancer and cardiovascular disease and generally occurs in favor of fission.

In a mouse model (FASEB J, 2021, Robert P ), the role of mitochondrial fusion has been demostrated as a protective factor against hypertension in resistance arteries and a deletion of OPA1 (optic Atrophy 1) fusion protein may lead to aneurysm until aortic dissection. The results of this experimental study suggest a role of the alteration of mitochondrial dynamic in the development of aneurysm and aortic dissection.

ELIGIBILITY:
Inclusion Criteria:

* Aneurysm aortic group: patients treated for an aneurysm of the ascending thoracic aorta with surgical indication according to the ESC guidelines (2014).
* Aortic dissection group: patients treated for type A acute aortic dissection or intramural hematoma of the ascending thoracic aorta in emergency.
* Control group: patients operated for aortic valve replacement (little aortic sample before closing aortotomy) or coronary artery bypass grafting which the use of a saphenous graft and the performance of a proximal anastomosis on the ascending aorta is planned

Exclusion Criteria:

* Patients under 18 years old
* Other acute aortic syndromes (penetrating ulcers, iatrogenic or traumatic dissections)
* Patients treated for aortic valve replacement in the context of infective endocarditis
* Patients treated for emergency aortic valve replacement or coronary bypass surgery**
* Pregnant, parturient and breastfeeding women
* Patients protected by an administrative or judicial measure (curatorship, guardianship)
* Patients receiving psychiatric care under duress
* Adults subject to a legal protection measure.
* Patients whose the samples planned for the study could not be taken;
* Patients in the control group whose tissue sampling will not be performed.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-09-07 (Actual); Primary Completion 2023-10-23 (Actual); Study Completion 2024-10-23 (Estimated)

PRIMARY OUTCOMES:
Level of tissue expression of the genes and coding for the proteins (Optic Atrophy 1) OPA1 | 1 month
  Level expression of, (Optic Atrophy 1) OPA1 by RT-qPCR
Level of tissue expression of the genes and coding for the proteins MFN1 (Mitofusin 1) | 1 month
  Level expression of MFN1 (Mitofusin 1) by RT-qPCR
Level of tissue expression of the genes and coding for the proteins MFN2 (Mitofusin 2) | 1 month
  Level expression of MFN2 (Mitofusin 2) by RT-qPCR
Level of tissue expression of the genes and coding for the proteins Fis1 | 1 month
  Level expression of Fis1 by RT-qPCR
Level of tissue expression of the genes and coding for the proteins Drp1 | 1 month
  Level expression of Drp1 by RT-qPCR
Level of tissue expression of the genes and coding for the proteins Nfr1 | 1 month
  Level expression of Nfr1 by RT-qPCR
Level of tissue expression of the genes and coding for the proteins Tfam | 1 month
  Level expression of Tfam by RT-qPCR
Level of tissue expression of the genes and coding for the proteins PGC1⍺ | 1 month
  Level expression of PGC1⍺ by RT-qPCR
Analysis of mitochondrial network | 1 month
  To analyze the mitochondrial network, vascular smooth muscle cells will be extracted from the wall of aorta samples and seeded in Petri dish. When 80% confluence is obtained, cells will be incubated with a green fluorescent marker (Mitotacker Green Probes) and 3D fluorescence microscopy will be used. Analysis of mitochondrial network will be done after characterization of mitochondrial shapes and distribution in the different aorta samples.

SECONDARY OUTCOMES:
Protein of remodelling and constitution of extracellular matrix: Metalloprotease MMp2 | 1 month
  Level expression of Metalloprotease MMp2 by western blot
Proteins of remodelling and constitution of extracellular matrix: Timp 1/2 | 1 month
  Level expression of Timp 1/2 by western blot
Proteins of remodelling and constitution of extracellular matrix: Collagene I/III | 1 month.
  Level expression of Collagene I/III by western blot
Protein of remodelling and constitution of extracellular matrix: Elastine | 1 month
  Level expression of Elastine by western blot
Proteins of survival cell: Bcl2/Bax | 1 month
  Level expression of Bcl2/Bax by western blot
Proteins of survival cell: Cytochrome C | 1 month
  Level expression of Cytochrome C by western blot
Proteins of oxydative stress: NADPH | 1 month
  Level expression of NADPH by western blot
Proteins of oxydative stress: OxyD | 1 month
  Level expression of OxyD by western blot
Proteins of oxydative stress: Sod 1/2 | 1 month
  Level expression of Sod 1/2 by western blot
Proteins of Smooth Muscle Cell reactivity: Myh11 | 1 month
  Level expression of Myh11 by western blot
Proteins of Smooth Muscle Cell reactivity: Acta 2 | 1 month
  Level expression of Acta 2 by western blot
Proteins of Smooth Muscle Cell reactivity: MLC20 | 1 month
  Level expression of MLC20 by western blot
Proteins of Smooth Muscle Cell reactivity: Rock1 | 1 month
  Level expression of Rock1 by western blot
Proteins of Smooth Muscle Cell reactivity: Rhoa | 1 month
  Level expression of Rhoa by western blot
Analysis of Plasma Metabolomes | 2 years
  154 metabolites will be measured in plasma samples. Plasma data blocks will be submitted to multiblock orthogonal component analysis (MOCA) after normalizing concentrations of plasma samples by their weights.
Analysis of Aorta Metabolomes | 2 years
  136 metabolites will be measured in plasma samples. Plasma data blocks will be submitted to multiblock orthogonal component analysis (MOCA) after normalizing concentrations of aorta samples by their weights.

CONTACTS AND LOCATIONS:
Locations (1):
- Olivier FOUQUET, Angers, France

IPD SHARING:
Plan to Share IPD: No
The data will be collected in a coded manner: first letter of the surname, first letter of the patient's first name, serial number of inclusion in the center by the physicians investigating the study in the electronic observation notebook managed by the DRCI of University Hospital of Angers

REFERENCES:
- [Background] Trabado S, Al-Salameh A, Croixmarie V, Masson P, Corruble E, Feve B, Colle R, Ripoll L, Walther B, Boursier-Neyret C, Werner E, Becquemont L, Chanson P. The human plasma-metabolome: Reference values in 800 French healthy volunteers; impact of cholesterol, gender and age. PLoS One. 2017 Mar 9;12(3):e0173615. doi: 10.1371/journal.pone.0173615. eCollection 2017. PMID 28278231
- [Result] Robert P, Nguyen PMC, Richard A, Grenier C, Chevrollier A, Munier M, Grimaud L, Proux C, Champin T, Lelievre E, Sarzi E, Vessieres E, Henni S, Prunier D, Reynier P, Lenaers G, Fassot C, Henrion D, Loufrani L. Protective role of the mitochondrial fusion protein OPA1 in hypertension. FASEB J. 2021 Jul;35(7):e21678. doi: 10.1096/fj.202000238RRR. PMID 34133045
- [Result] Toda M, Yamamoto K, Shimizu N, Obi S, Kumagaya S, Igarashi T, Kamiya A, Ando J. Differential gene responses in endothelial cells exposed to a combination of shear stress and cyclic stretch. J Biotechnol. 2008 Jan 20;133(2):239-44. doi: 10.1016/j.jbiotec.2007.08.009. Epub 2007 Aug 9. PMID 17850909
- [Result] Archer SL. Mitochondrial dynamics--mitochondrial fission and fusion in human diseases. N Engl J Med. 2013 Dec 5;369(23):2236-51. doi: 10.1056/NEJMra1215233. No abstract available. PMID 24304053
- [Result] Piquereau J, Caffin F, Novotova M, Prola A, Garnier A, Mateo P, Fortin D, Huynh le H, Nicolas V, Alavi MV, Brenner C, Ventura-Clapier R, Veksler V, Joubert F. Down-regulation of OPA1 alters mouse mitochondrial morphology, PTP function, and cardiac adaptation to pressure overload. Cardiovasc Res. 2012 Jun 1;94(3):408-17. doi: 10.1093/cvr/cvs117. Epub 2012 Mar 8. PMID 22406748
- [Result] Le Page S, Niro M, Fauconnier J, Cellier L, Tamareille S, Gharib A, Chevrollier A, Loufrani L, Grenier C, Kamel R, Sarzi E, Lacampagne A, Ovize M, Henrion D, Reynier P, Lenaers G, Mirebeau-Prunier D, Prunier F. Increase in Cardiac Ischemia-Reperfusion Injuries in Opa1+/- Mouse Model. PLoS One. 2016 Oct 10;11(10):e0164066. doi: 10.1371/journal.pone.0164066. eCollection 2016. PMID 27723783